CLINICAL TRIAL: NCT04419103
Title: Study on Physiologic Requirement and Dietary Recommended Nutrient
Brief Title: Study on Physiologic Requirement and Dietary Recommended Nutrient Intake (RNI) of Iodine in Children
Status: Completed | Type: Observational
Sponsor: Tianjin Medical University (Other)
Collaborators: Shandong Institute for Endemic Disease Control and Research (Unknown)
Responsible Party: Principal Investigator, Chen Wen, Teacher, Tianjin Medical University
Other Study IDs: NSFC-81803223
Record Dates: First submitted 2020-06-01; First posted 2020-06-05 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Nutritional Requirements
Keywords: nutrient; public nutrition; nutrition related diseases; nutrition epidemiology

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — 1. Iodine nutrition survey of children was carried out in the villages and towns with low water iodine and no iodized salt supply. Basic information, venous blood, water samples, dietary information, spot urine and two 24-hour (24-h) urine were collected and thyroid ultrasound was performed to comprehensively assess children's thyroid function and iodine nutrition status. 2. An iodine balance experiment was conducted in children. All food and water ingested by the subjects were measured by the weighing method, and 24-h urine and feces were collected. Iodine intake and excretion were assessed, and saliva samples were collected six times a day.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — Natural exposure of iodine.

SUMMARY:
Iodine is one of essential micronutrient for human, both iodine deficiency and excess will be harmful for human health. Children is the susceptible population to iodine nutrition, and studies show that even mild iodine deficiency would affect the growth and development of children, so it is urgent to identify the dietary recommended nutrient intake (RNI) of iodine for children to guide children scientifically and safely supplement iodine. There are few studies about the dietary recommended nutrient intake (RNI) of iodine in children, and present data are old and outdated.

DETAILED DESCRIPTION:
Based on the investigators'previous study on upper safe level of iodine on children from areas with high iodine in drinking water, this study will conduct an epidemiological study on 600 children living in areas with high water iodine content but the actual iodine content in participants' drinking water is not so high, while no supply of iodized salt.

Meanwhile, in order to get iodine dietary recommended nutrient intake (RNI) values of children. The investigators will conduct a iodine balance experiment on children with sufficient iodine nutrition. We will randomly select thirty healthy students for a three-day iodine balance experiment from the cross-sectional study. The investigators will use the regression model to obtain an iodine intake value when children at"zero iodine"balance. Combine the study at population and individual level, the investigators will obtain data on dietary recommended nutrient intake (RNI) of iodine for Chinese children, to properly guide children iodine supplementation to avoid iodine deficiency, which also will provide data for the update of Chinese dietary reference intakes of iodine.

ELIGIBILITY:
Inclusion Criteria:

Normal body mass index and thyroid function have not been treated for thyroid disease have not used amiodarone and other drugs (including iodine supplements) during the investigation have no major diseases and family history have lived in the local area for more than 5 years

Exclusion Criteria:

Long-term low-protein long-term low-heat energy malnutrition

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 7-11 years old Primary school students who in grades 2, 3, 4 and 5 are the research subjects.They were recruited in Shandong.
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
urinary iodine concentration | 2 weeks
  μg/L
free triiodothyronine | 2 weeks
  pmol/L
water iodine intake | 2 weeks
  μg/day
diet iodine intake | 2 weeks
  μg/day
salt iodine concentration | 2 weeks
  μg/L
free thyroxine | 2 weeks
  pmol/L
thyroid-stimulating hormone | 2 weeks
  mIU/L
thyroperoxidase antibody | 2 weeks
  IU/mL
thyroglobulin antibody | 2 weeks
  IU/mL
urinary iodine excretion | 2 weeks
  μg/day
fecal iodine excretion | 2 weeks
  μg/day

CONTACTS AND LOCATIONS:
Overall Officials: xiao ming Wang, Principal Investigator — Shandong Institute for Endemic Disease Control and Research; gui jun Tan, Principal Investigator — The First Central Hospital of Tianjin Medical University; man Zhang, Principal Investigator — Shandong Institute for Endemic Disease Control and Research
Locations (1):
- Shandong Institute for Endemic Disease Control and Research, Dezhou, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sang Z, Chen W, Shen J, Tan L, Zhao N, Liu H, Wen S, Wei W, Zhang G, Zhang W. Long-term exposure to excessive iodine from water is associated with thyroid dysfunction in children. J Nutr. 2013 Dec;143(12):2038-43. doi: 10.3945/jn.113.179135. Epub 2013 Oct 9. PMID 24108132
- [Background] Brantsaeter AL, Knutsen HK, Johansen NC, Nyheim KA, Erlund I, Meltzer HM, Henjum S. Inadequate Iodine Intake in Population Groups Defined by Age, Life Stage and Vegetarian Dietary Practice in a Norwegian Convenience Sample. Nutrients. 2018 Feb 17;10(2):230. doi: 10.3390/nu10020230. PMID 29462974
- [Background] Pal N, Samanta SK, Chakraborty A, Chandra NK, Chandra AK. Interrelationship between iodine nutritional status of lactating mothers and their absolutely breast-fed infants in coastal districts of Gangetic West Bengal in India. Eur J Pediatr. 2018 Jan;177(1):39-45. doi: 10.1007/s00431-017-3025-6. Epub 2017 Oct 23. PMID 29063209
- [Background] Zimmermann MB, Andersson M. Update on iodine status worldwide. Curr Opin Endocrinol Diabetes Obes. 2012 Oct;19(5):382-7. doi: 10.1097/MED.0b013e328357271a. PMID 22892867
- [Background] Delshad H, Mirmiran P, Abdollahi Z, Salehi F, Azizi F. Continuously sustained elimination of iodine deficiency: a quarter of a century success in the Islamic Republic of Iran. J Endocrinol Invest. 2018 Sep;41(9):1089-1095. doi: 10.1007/s40618-018-0838-8. Epub 2018 Feb 14. PMID 29446011
- [Background] Andersson M, Karumbunathan V, Zimmermann MB. Global iodine status in 2011 and trends over the past decade. J Nutr. 2012 Apr;142(4):744-50. doi: 10.3945/jn.111.149393. Epub 2012 Feb 29. PMID 22378324
- [Background] Murcia M, Espada M, Julvez J, Llop S, Lopez-Espinosa MJ, Vioque J, Basterrechea M, Riano I, Gonzalez L, Alvarez-Pedrerol M, Tardon A, Ibarluzea J, Rebagliato M. Iodine intake from supplements and diet during pregnancy and child cognitive and motor development: the INMA Mother and Child Cohort Study. J Epidemiol Community Health. 2018 Mar;72(3):216-222. doi: 10.1136/jech-2017-209830. Epub 2017 Dec 26. PMID 29279360
- [Background] Zimmermann MB, Ito Y, Hess SY, Fujieda K, Molinari L. High thyroid volume in children with excess dietary iodine intakes. Am J Clin Nutr. 2005 Apr;81(4):840-4. doi: 10.1093/ajcn/81.4.840. PMID 15817861
- [Background] Chen W, Li X, Wu Y, Bian J, Shen J, Jiang W, Tan L, Wang X, Wang W, Pearce EN, Zimmermann MB, Carriquiry AL, Zhang W. Associations between iodine intake, thyroid volume, and goiter rate in school-aged Chinese children from areas with high iodine drinking water concentrations. Am J Clin Nutr. 2017 Jan;105(1):228-233. doi: 10.3945/ajcn.116.139725. Epub 2016 Dec 7. PMID 27927635
- [Background] Aakre I, Strand TA, Moubarek K, Barikmo I, Henjum S. Associations between thyroid dysfunction and developmental status in children with excessive iodine status. PLoS One. 2017 Nov 22;12(11):e0187241. doi: 10.1371/journal.pone.0187241. eCollection 2017. PMID 29166388
- [Background] Calza L, Fernandez M, Giardino L. Cellular approaches to central nervous system remyelination stimulation: thyroid hormone to promote myelin repair via endogenous stem and precursor cells. J Mol Endocrinol. 2010 Jan;44(1):13-23. doi: 10.1677/JME-09-0067. Epub 2009 Jul 3. PMID 19578096
- [Background] Liu HL, Lam LT, Zeng Q, Han SQ, Fu G, Hou CC. Effects of drinking water with high iodine concentration on the intelligence of children in Tianjin, China. J Public Health (Oxf). 2009 Mar;31(1):32-8. doi: 10.1093/pubmed/fdn097. Epub 2008 Oct 23. PMID 18952598
- [Background] Malvaux P, Beckers C, De Visscher M. Iodine balance studies in nongoitrous children and in adolescents on low iodine intake. J Clin Endocrinol Metab. 1969 Jan;29(1):79-84. doi: 10.1210/jcem-29-1-79. No abstract available. PMID 5762324
- [Background] Sang Z, Wang PP, Yao Z, Shen J, Halfyard B, Tan L, Zhao N, Wu Y, Gao S, Tan J, Liu J, Chen Z, Zhang W. Exploration of the safe upper level of iodine intake in euthyroid Chinese adults: a randomized double-blind trial. Am J Clin Nutr. 2012 Feb;95(2):367-73. doi: 10.3945/ajcn.111.028001. Epub 2011 Dec 28. PMID 22205314
- [Background] Pearce EN, Andersson M, Zimmermann MB. Global iodine nutrition: Where do we stand in 2013? Thyroid. 2013 May;23(5):523-8. doi: 10.1089/thy.2013.0128. Epub 2013 Apr 18. PMID 23472655
- [Background] Mason JB, Deitchler M, Gilman A, Gillenwater K, Shuaib M, Hotchkiss D, Mason K, Mock N, Sethuraman K. Iodine fortification is related to increased weight-for-age and birthweight in children in Asia. Food Nutr Bull. 2002 Sep;23(3):292-308. doi: 10.1177/156482650202300309. PMID 12362593
- [Background] Zimmermann MB, Jooste PL, Mabapa NS, Mbhenyane X, Schoeman S, Biebinger R, Chaouki N, Bozo M, Grimci L, Bridson J. Treatment of iodine deficiency in school-age children increases insulin-like growth factor (IGF)-I and IGF binding protein-3 concentrations and improves somatic growth. J Clin Endocrinol Metab. 2007 Feb;92(2):437-42. doi: 10.1210/jc.2006-1901. Epub 2006 Nov 21. PMID 17118996
- [Background] Hynes KL, Otahal P, Hay I, Burgess JR. Mild iodine deficiency during pregnancy is associated with reduced educational outcomes in the offspring: 9-year follow-up of the gestational iodine cohort. J Clin Endocrinol Metab. 2013 May;98(5):1954-62. doi: 10.1210/jc.2012-4249. Epub 2013 Apr 30. PMID 23633204
- [Background] Hynes KL, Otahal P, Burgess JR, Oddy WH, Hay I. Reduced Educational Outcomes Persist into Adolescence Following Mild Iodine Deficiency in Utero, Despite Adequacy in Childhood: 15-Year Follow-Up of the Gestational Iodine Cohort Investigating Auditory Processing Speed and Working Memory. Nutrients. 2017 Dec 13;9(12):1354. doi: 10.3390/nu9121354. PMID 29236073
- [Background] Vannucchi G, Covelli D, Vigo B, Perrino M, Mondina L, Fugazzola L. Thyroid volume and serum calcitonin changes during pregnancy. J Endocrinol Invest. 2017 Jul;40(7):727-732. doi: 10.1007/s40618-017-0622-1. Epub 2017 Feb 22. PMID 28229359
- [Background] Lazarus JH. Thyroid function in pregnancy. Br Med Bull. 2011;97:137-48. doi: 10.1093/bmb/ldq039. Epub 2010 Dec 23. PMID 21186204
- [Derived] Guo W, Yang Y, Jiang W, Cheng Y, Wu W, Pan Z, Zhang D, Li S, Ren Z, Zhang N, Zhang K, Pearce EN, Chen W, Zhang W. An Iodine Balance Study in Chinese School-age Children. J Clin Endocrinol Metab. 2023 Sep 18;108(10):e949-e955. doi: 10.1210/clinem/dgad244. PMID 37146180
- [Derived] Guo W, Pan Z, Zhang Y, Jin Y, Dong S, Wu W, Chen W, Zhang W. Saliva Iodine Concentration in Children and Its Association with Iodine Status and Thyroid Function. J Clin Endocrinol Metab. 2020 Sep 1;105(9):dgaa471. doi: 10.1210/clinem/dgaa471. PMID 32687189